CLINICAL TRIAL: NCT04463641
Title: Assessment of the Axone Micro Quadripolar Lead for Enhanced Cardiac Resynchronization Therapy
Acronym: ASTRAL-4LV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAXI01
Record Dates: First submitted 2020-06-23; First posted 2020-07-09 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy
Keywords: Left Ventricular Lead
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Axone 4LV Lead (Experimental): Subjects implanted with the Axone 4LV Lead
  Interventions: Device: Implantation of the Axone 4LV Lead

INTERVENTIONS:
Device: Implantation of the Axone 4LV Lead — Implantation of the Axone 4LV Lead

SUMMARY:
The primary objective of this study is to assess the chronic safety and performance of the Axone left ventricular (LV) micro-lead.

DETAILED DESCRIPTION:
This is a interventional, pivotal, prospective, single arm, open label, multicenter, international trial.

The device under investigation is the Axone system, consisting of:

* Axone 4LV: an ultrathin, lumenless, quadripolar, IS4-compatible lead designed for left ventricular pacing for cardiac resynchronization therapy (CRT).
* Axone µGuide: a dedicated, permanently implantable micro catheter designed for implantation of the Axone 4LV lead.

The primary endpoint data will be used to support CE marking of the Axone system.

The primary endpoints will be evaluated at 6 months post-implantation. Subjects will be followed-up at 6 weeks, 3 months, 6 months, 12 months post-implantation, then yearly until 4 years post-implantation.

ELIGIBILITY:
Inclusion Criteria:

* Indication for cardiac resynchronization therapy-defibrillator (CRT-D) device implant according to the latest ESC (European Society of Cardiology) guidelines
* De-novo implant of a Platinium 4LV CRT-D device (or any newer 4LV CRT-D model manufactured by MicroPort CRM)
* Reviewed, signed and dated informed consent form

Exclusion Criteria:

* LV lead previous implant attempt
* Upgrade to CRT from a previously implanted pacemaker or implantable cardioverter-defibrillator (ICD), or CRT device replacement
* Known allergy to contrast media used for imaging during cardiac catheterization
* Tricuspid valvular disease or any type of tricuspid replacement heart valve (mechanical or tissue)
* Severe renal failure (creatinine clearance according to the Modification of Diet in Renal Disease (MDRD) formula < 30ml/min/m²)
* Active myocarditis
* Stroke, myocardial infarction or cardiac revascularization within 40 days prior to implant
* Previous heart transplant or currently on heart transplant list
* Life expectancy less than 1 year
* Already included in another clinical study that could confound the results of this study
* Pre-menopausal women / women in childbearing age, including pregnant and breastfeeding women
* Less than 18 years old or under guardianship
* Incapacitated subject, inability to understand the purpose of the study, or to meet follow-up visits at the implanting site as defined in the protocol
* Diagnosis of drug addiction (substance use disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety co-primary endpoint, defined as Axone system related complication free rate at 6 months post implant | 6 months
  A complication is defined as any Serious Adverse Device Effect (SADE) resulting in death or requiring invasive intervention. Safety co-primary endpoint assessment will be based on independent event adjudication by a Clinical Event Committee (CEC).
Performance co-primary endpoint, defined as LV pacing success rate at 6 months post implant | 6 months
  LV pacing success is defined as at least one LV pacing vector with:
  * Pacing Threshold (PT) ≤ 3.5V at 1ms pulse width, and
  * No phrenic nerve stimulation at PT+2V / 1ms pulse width.

SECONDARY OUTCOMES:
Bizone LV pacing success rate at 6 months post implant | 6 months
  Bizone LV pacing success is defined as two distant pacing vectors with:
  * A Pacing Threshold (PT) ≤ 3.5V at 1ms pulse width, and
  * No phrenic nerve stimulation at PT +2V / 1ms pulse width. Two pacing vectors are considered distant when cathode electrodes are separated by at least 30 mm.

OTHER OUTCOMES:
Axone 4LV implantation success rate | At implant, preferably within 15 days of enrollment
Implantation duration | At implant, preferably within 15 days of enrollment
Fluoroscopy time | At implant, preferably within 15 days of enrollment
  Fluoroscopy time is measured in minutes
Fluoroscopy dose | At implant, preferably within 15 days of enrollment
  Fluoroscopy dose is measured using dose area product (Gray.cm^2)
Axone system handling assessment | At implant, preferably within 15 days of enrollment
  Implanters will be asked to fill in a handling questionnaire and record observations related to the use of the Axone system.
Axone implanters' learning curve | At implant, preferably within 15 days of enrollment
  This endpoint will be based on fluoroscopy time for implantation. The effect of removing the 1st, 2nd, 3rd, etc implanted subjects on mean fluoroscopy time (per implanter and per site) will be calculated.
Number of excitable myocardium areas at implant | At implant, preferably within 15 days of enrollment
  "Excitable myocardium areas" are areas that can be paced by the implanted Axone 4LV lead.
Effect of CRT therapy, in particular bizone pacing, on QRS parameters, at discharge and 6 months post implant | At discharge, within 7 days of implant, and at 6 months
  The effect of monozone and bizone CRT pacing on duration of QRS is measured in milliseconds.
Effect of CRT therapy, in particular bizone pacing, on Left Pre-Ejection Interval (LPEI), at discharge | At discharge, within 7 days of implant
  LPEI (in milliseconds) is an electromechanical parameter that can be assessed using echocardiography.
Axone 4LV lead pacing threshold | Discharge (within 7 days of implant), 6 weeks, 3 months, 6 months, 12 months, 24 months 36 months, 48 months
  Pacing threshold is measured in Volts.
Axone 4LV lead pacing impedance | Discharge (within 7 days of implant), 6 weeks, 3 months, 6 months, 12 months, 24 months 36 months, 48 months
  Pacing impedance is measured in Ohms.
Presence of phrenic nerve stimulation (PNS) with the Axone 4LV lead | Implant (preferably within 15 days of enrollment), discharge (within 7 days of implant), 6 weeks, 3 months, 6 months
  The presence of PNS will be assessed at 10V using an external pacing system analyzer at implant, or at pacing threshold +2V at other visits.
Axone 4LV lead programming | Discharge (within 7 days of implant), 6 weeks, 3 months, 6 months, 12 months, 24 months 36 months, 48 months
  Lead programming will be reported using: (i) pacing amplitude (Volts), pulse width (milliseconds) and pacing vector(s) selected.
Energy consumption associated with Axone 4LV lead | 6 months
  Energy will be calculated using the formula: E=(pacing amplitude^2 x pulse width)/impedance. Energy, pacing amplitude, pulse width and impedance are measured in Joules, Volts, milliseconds, and Ohms, respectively.
Axone system-related annual complication-free rate | 12 months, 24 months 36 months, 48 months
  Definition of Axone system related complication is the same as for primary safety endpoint.
Clinical response to CRT at 12 months post implant | 12 months
  Clinical response will be determined by looking at functional improvement, reverse remodelling, freedom from heart failure events, and rate of non-responders:
  (i) functional improvement is defined as improvement in ≥1 NYHA (New York Heart Association) class from baseline to 12 months.
  (ii) reverse remodelling is a ≥12% increase in left ventricular end systolic volume index (LVESVi: LVESV [mL] and body surface area [m^2] will be combined to report LVESVi).
  (iii) freedom from heart failure events is defined as an absence of death or HF hospitalization.
  (iv) non-responders are all those who are not responders. A responder is defined as a subject that is not dead and who did not experience any HF hospitalization and that has a stable or improved NYHA class versus baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Anselme, MD, Principal Investigator — CHU de Rouen, France
Locations (21):
- Kepler Universitätsklinikum, Linz, Austria
- France (8):
  - CH Annecy Genevois, Annecy
  - CHRU Hopital Trousseau, Chambray-lès-Tours
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHRU de Lille - Hôpital Cardiologique, Lille
  - CHU Pontchaillou, Rennes
  - CHU de Rouen, Rouen
  - CHU Toulouse, Toulouse
- Germany (3):
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
- Italy (3):
  - ASST Spedali Civili di Brescia, Brescia
  - Ospedale Pellegrini, Naples
  - Ospedale Policlinico Federico II, Naples
- Isala Klinieken, Zwolle, Netherlands
- Portugal (2):
  - Centro Hospitalar Universitário Lisboa Norte - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Universitário do Porto, Porto
- Spain (3):
  - Hospital Universitario General de Alicante, Alicante
  - Hospital Universitario La Fe, Valencia
  - Hospital Álvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] Linde C, Abraham WT, Gold MR, St John Sutton M, Ghio S, Daubert C; REVERSE (REsynchronization reVErses Remodeling in Systolic left vEntricular dysfunction) Study Group. Randomized trial of cardiac resynchronization in mildly symptomatic heart failure patients and in asymptomatic patients with left ventricular dysfunction and previous heart failure symptoms. J Am Coll Cardiol. 2008 Dec 2;52(23):1834-1843. doi: 10.1016/j.jacc.2008.08.027. Epub 2008 Nov 7. PMID 19038680
- [Background] Zeitler EP, Friedman DJ, Daubert JP, Al-Khatib SM, Solomon SD, Biton Y, McNitt S, Zareba W, Moss AJ, Kutyifa V. Multiple Comorbidities and Response to Cardiac Resynchronization Therapy: MADIT-CRT Long-Term Follow-Up. J Am Coll Cardiol. 2017 May 16;69(19):2369-2379. doi: 10.1016/j.jacc.2017.03.531. PMID 28494974
- [Background] Healey JS, Hohnloser SH, Exner DV, Birnie DH, Parkash R, Connolly SJ, Krahn AD, Simpson CS, Thibault B, Basta M, Philippon F, Dorian P, Nair GM, Sivakumaran S, Yetisir E, Wells GA, Tang AS; RAFT Investigators. Cardiac resynchronization therapy in patients with permanent atrial fibrillation: results from the Resynchronization for Ambulatory Heart Failure Trial (RAFT). Circ Heart Fail. 2012 Sep 1;5(5):566-70. doi: 10.1161/CIRCHEARTFAILURE.112.968867. Epub 2012 Aug 14. PMID 22896584
- [Background] Daubert C, Behar N, Martins RP, Mabo P, Leclercq C. Avoiding non-responders to cardiac resynchronization therapy: a practical guide. Eur Heart J. 2017 May 14;38(19):1463-1472. doi: 10.1093/eurheartj/ehw270. PMID 27371720
- [Background] Okamura H. Up-to-date cardiac resynchronization therapy. J Gen Fam Med. 2017 May 17;18(5):195-199. doi: 10.1002/jgf2.24. eCollection 2017 Oct. PMID 29264026
- [Background] Macias A, Gavira JJ, Alegria E, Azcarate PM, Barba J, Garcia-Bolao I. [Effect of the left ventricular pacing site on echocardiographic parameters of ventricular dyssynchrony in patients receiving cardiac resynchronization therapy]. Rev Esp Cardiol. 2004 Feb;57(2):138-45. Spanish. PMID 14967109
- [Background] Butter C, Auricchio A, Stellbrink C, Fleck E, Ding J, Yu Y, Huvelle E, Spinelli J; Pacing Therapy for Chronic Heart Failure II Study Group. Effect of resynchronization therapy stimulation site on the systolic function of heart failure patients. Circulation. 2001 Dec 18;104(25):3026-9. doi: 10.1161/hc5001.102229. PMID 11748094
- [Background] Umar F, Taylor RJ, Stegemann B, Marshall H, Flannigan S, Lencioni M, De Bono J, Griffith M, Leyva F. Haemodynamic effects of cardiac resynchronization therapy using single-vein, three-pole, multipoint left ventricular pacing in patients with ischaemic cardiomyopathy and a left ventricular free wall scar: the MAESTRO study. Europace. 2016 Aug;18(8):1227-34. doi: 10.1093/europace/euv396. Epub 2015 Dec 30. PMID 26718535
- [Background] Bonadei I, Vizzardi E, Gorga E, Carubelli V, Pagnoni M, Sciatti E, Raweh A, Cerini M, Bontempi L, Curnis A, Metra M. Role of the old and new echocardiographic technologies in cardiac resynchronization therapy. Minerva Cardioangiol. 2016 Oct;64(5):572-80. Epub 2015 Jun 23. PMID 26099222
- [Background] O'Brien T, Park MS, Youn JC, Chung ES. The Past, Present and Future of Cardiac Resynchronization Therapy. Korean Circ J. 2019 May;49(5):384-399. doi: 10.4070/kcj.2019.0114. PMID 31074211
- [Background] Leclercq C, Burri H, Curnis A, Delnoy PP, Rinaldi CA, Sperzel J, Lee K, Calo L, Vicentini A, Concha JF, Thibault B. Cardiac resynchronization therapy non-responder to responder conversion rate in the more response to cardiac resynchronization therapy with MultiPoint Pacing (MORE-CRT MPP) study: results from Phase I. Eur Heart J. 2019 Sep 14;40(35):2979-2987. doi: 10.1093/eurheartj/ehz109. PMID 30859220
- [Background] Auricchio A, Heggermont WA. Technology Advances to Improve Response to Cardiac Resynchronization Therapy: What Clinicians Should Know. Rev Esp Cardiol (Engl Ed). 2018 Jun;71(6):477-484. doi: 10.1016/j.rec.2018.01.006. Epub 2018 Feb 14. English, Spanish. PMID 29454549
- [Background] Antoniadis AP, Behar JM, Sieniewicz B, Gould J, Niederer S, Rinaldi CA. A comparison of the different features of quadripolar left ventricular pacing leads to deliver cardiac resynchronization therapy. Expert Rev Med Devices. 2017 Sep;14(9):697-706. doi: 10.1080/17434440.2017.1369404. Epub 2017 Aug 23. PMID 28835138
- [Background] Tomassoni G, Baker J, Corbisiero R, Love C, Martin D, Niazi I, Sheppard R, Worley S, Beau S, Greer GS, Aryana A, Cao M, Harbert N, Zhang S; Promote(R) Q CRT-D and Quartet(R) Left Ventricular Heart Lead Study Group. Postoperative performance of the Quartet(R) left ventricular heart lead. J Cardiovasc Electrophysiol. 2013 Apr;24(4):449-56. doi: 10.1111/jce.12065. Epub 2013 Jan 22. PMID 23339555
- [Background] Crossley GH, Biffi M, Johnson B, Lin A, Gras D, Hussin A, Cuffio A, Collier JL, El-Chami M, Li S, Holloman K, Exner DV. Performance of a novel left ventricular lead with short bipolar spacing for cardiac resynchronization therapy: primary results of the Attain Performa quadripolar left ventricular lead study. Heart Rhythm. 2015 Apr;12(4):751-8. doi: 10.1016/j.hrthm.2014.12.019. Epub 2014 Dec 19. PMID 25533587
- [Background] Mittal S, Nair D, Padanilam BJ, Ciuffo A, Gupta N, Gallagher P, Goldner B, Hammill EF, Wold N, Stein K, Burke M. Performance of Anatomically Designed Quadripolar Left Ventricular Leads: Results from the NAVIGATE X4 Clinical Trial. J Cardiovasc Electrophysiol. 2016 Oct;27(10):1199-1205. doi: 10.1111/jce.13044. Epub 2016 Aug 19. PMID 27434039